CLINICAL TRIAL: NCT00461227
Title: Genes, Home Allergens, and Asthma in Puerto Rican Children
Brief Title: Effect of Heredity and Environment on Asthma Development and Severity in Puerto Rican Children
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Juan Celedon, MD, Professor of Pediatrics, University of Pittsburgh
Other Study IDs: 1353; R01HL079966-01A2 (NIH)
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Asthma; Hypersensitivity
Keywords: Puerto Rican; Allergies
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma is a major public health problem among Puerto Ricans. Little is known, however, about the effect of heredity and environment on the development and severity of asthma in this population. This study will examine the relationship between asthma and certain genetic and environmental factors in Puerto Rican children.

DETAILED DESCRIPTION:
Asthma is a chronic disease that causes constriction of the airways. People with asthma may experience wheezing, coughing, chest tightness, and trouble breathing. Although asthma is a major public health problem among Puerto Ricans, little research has been done to determine the influence of heredity and environment on the disease in this population. To learn more about these relationships, this study will examine the effects of certain genes and allergens on the development and severity of asthma in Puerto Rican children.

This observational study will recruit both children with asthma and children without asthma. Participants will meet with study staff twice during the study. The first visit will take place at participants' homes. Participants will complete questionnaires about demographics, respiratory and general health, and household characteristics. Lung function testing, collection of blood samples, and collection of household dust samples will also take place at the home-based visit. The second visit will take place at the study site. At this visit, participants will undergo allergy tests on the skin and a methacholine challenge test to assess their airway responsiveness and asthma severity. The methacholine challenge test will involve inhaling mist through a mouthpiece and blowing forcefully into a special apparatus called a spirometer. Parents will be asked to provide information about their children's exposure to pets in early life. Each visit will last approximately 1.5 hours and will be scheduled close to the date on which a participant enters the study.

ELIGIBILITY:
Inclusion Criteria:

For participants with asthma:

* Diagnosis of asthma
* History of wheezing within 12 months prior to study entry
* Has four grandparents that were born in Puerto Rico

For participants without asthma:

* No diagnosis of asthma
* No history of wheezing within 12 months prior to study entry
* Has four grandparents that were born in Puerto Rico

Exclusion Criteria:

* Significant pulmonary disease other than asthma
* Hospitalization in the neonatal intensive care unit and requiring ventilatory support
* History of cigarette smoking for more than 5 pack-years ([number of packs smoked per day] x [number of years of smoking])

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children of Puerto Rican descent (having four Puerto Rican grandparents) living in Hartford (Connecticut) and in the metropolitan areas of San Juan and Caguas in the island of Puerto Rico.
Sampling Method: Probability Sample
Enrollment: 1127 (Actual)
Dates: Start 2006-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Effect of certain genes and allergens on the development and severity of asthma in Puerto Rican children | Measured at participants' two study visits

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Celedon, MD, DrPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- University of Puerto Rico, San Juan, Puerto Rico